CLINICAL TRIAL: NCT03342638
Title: Maximizing Outcome of Multiple Sclerosis Transplantation: "MOST" Trial
Brief Title: Maximizing Outcome of Multiple Sclerosis Transplantation
Acronym: MOST
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: PI Sabbatical
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richard Burt, MD, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIAD.MOST.2017
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Results first posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Autologous Stem Cell Transplantation; Stem Cells; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Cyclophosphamide; Mesna; thymoglobulin; Methylprednisolone; Methylprednisolone Hemisuccinate; Granulocyte Colony-Stimulating Factor; Filgrastim; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (Experimental): Hematopoietic Stem Cell Therapy will be performed as follows: Autologous stem cells will be infused after conditioning with cyclophosphamide, mesna, rATG (rabbit), and methylprednisolone. Granulocyte-colony stimulating factor (G-CSF) will be administered post-transplant.
  Interventions: Drug: Cyclophosphamide; Drug: Mesna; Drug: rATG; Drug: Methylprednisolone; Drug: G-CSF; Biological: Autologous Stem Cells
- IVIg Arm (Experimental): Hematopoietic Stem Cell Therapy will be performed as follows: Autologous stem cells will be infused after conditioning with cyclophosphamide, mesna, rATG (rabbit), and methylprednisolone. IVIg and G-CSF will be administered post-transplant.
  Interventions: Drug: Cyclophosphamide; Drug: Mesna; Drug: rATG; Drug: Methylprednisolone; Drug: G-CSF; Biological: IVIg; Biological: Autologous Stem Cells

INTERVENTIONS:
Drug: Cyclophosphamide — Potent immunosuppressive agent; an alkylating agent
  Other Names: Cytoxan; Neosar
Drug: Mesna — Medication used to decrease the risk of hemorrhagic cystitis prophylaxis
  Other Names: Mesnex
Drug: rATG — A predominantly lymphocyte-specific immunosuppressive agent which contains antibodies specific to the antigens commonly found on the surface of T cells
  Other Names: Thymoglobulin
Drug: Methylprednisolone — Steroid
  Other Names: Solu-Medrol
Drug: G-CSF — Granulocyte-colony stimulating factor; a glycoprotein that stimulates the bone marrow to produce granulocytes and stem cells and release them into the bloodstream
  Other Names: Neupogen; Filgrastim; Granix; Zarxio
Biological: IVIg — Sterile, purified immunoglobulin G (IgG) products manufactured from pooled human plasma and typically contain more than 95% unmodified IgG, which has intact Fc-dependent effector functions and only trace amounts of immunoglobulin A (IgA) or immunoglobulin M (IgM).
  Other Names: Gammagard; Carimune Nanofiltered (NF); Bivagam; Privigen
  Arms: IVIg Arm
Biological: Autologous Stem Cells — Infusion of participant's own stem cells

SUMMARY:
Randomized study of autologous un-manipulated peripheral blood hematopoietic stem cell transplant (HSCT) comparing two regimens: (1) cyclophosphamide and rabbit anti-thymoglobulin (rATG) versus (2) cyclophosphamide, rATG, and Intravenous Immunoglobulin (IVIg).

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is at onset an immune-mediated demyelinating disease. In most cases, it starts as a relapsing-remitting disease with distinct attacks and no symptoms between flares. Over years or decades, virtually all cases transition into a progressive disease in which insidious and slow neurologic deterioration occurs with or without acute flares. Relapsing-remitting disease is often responsive to immune suppressive or modulating therapies, while immune based therapies are generally ineffective in patients with a progressive clinical course. This clinical course and response to immune suppression, as well as neuropathology and neuroimaging studies, suggest that disease progression is associated with axonal atrophy. Disability correlates better with measures of axonal atrophy than immune mediated demyelination. Therefore, immune based therapies, in order to be effective, need to be started early in the disease course while MS is predominantly an immune-mediated and inflammatory disease. While current immune based therapies delay disability, no intervention has been proven to prevent progressive disability.The investigators propose a randomized study of autologous unmanipulated peripheral blood hematopoietic stem cell transplant (HSCT) comparing two different conditioning regimens: (1) cyclophosphamide and rabbit anti-thymoglobulin (rATG) versus (2) cyclophosphamide, rATG, and Intravenous Immunoglobulin (IVIg).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-58 years
2. Diagnosis of MS using revised McDonald criteria of clinically definite MS (Appendix A)
3. An EDSS score of 2.0 to 6.0 (Appendix B).
4. An EDSS >6.0 may be included if still relapsing-remitting disease and at least two enhancing lesions on MRI within the last three months
5. Inflammatory disease despite treatment with standard disease modifying therapy (DMT) including at least 6 months of interferon or Copaxone. Inflammatory disease is defined based on either MRI (gadolinium enhancing lesion, new T2 lesion) or *steroid-treated clinical relapses (prescribed by a neurologist)
6. Minimum disease activity required:

   1. Failed a first line DMT (Copaxone or Interferon), defined as two or more *steroid treated clinical relapses within the last 12 months. A clinical relapse may also be evidence of active inflammation on MRI (gadolinium enhancing lesion or new T2 lesion) in the last 12 months on two MRIs at least three months apart
   2. Failed a second or third line MS Drug: Zinbryta (daclizumab), Aubagio (teriflunomide), Gilenya (fingolimod), Tecifidera (dimethyl fumarate), Lemtrada (alemtuzumab), Ocrevus (ocrelizumab), Tysabri (natalizumab), Rituxan (rituximab) or IVIg, defined as one *steroid treated clinical relapse within the last 12 months or evidence of active inflammation on MRI (gadolinium enhancing lesion or new T2 lesion) in the last 12 months.
   3. Cognitive dysfunction that prevents gainful employment, but competent to comply with treatment and informed consent

      * A steroid-treated relapse will include a relapse that was severe enough to justify treatment but due to patient intolerance of steroids, they were offered but not used.

Exclusion Criteria:

1. Any adult who is unable to consent (for adults who are cognitively impaired due to MS, consent may be obtained from the closest living relative or person who has power of attorney)
2. Individuals under the age of 18 or over the age of 58
3. Diagnosis of Primary Progressive MS, Secondary Progressive MS, or Clinically Isolated Syndrome (CIS)
4. Pregnant women (positive serum or urine human chorionic gonadotropin (HCG) test)
5. Women who are breastfeeding
6. Prisoners
7. Any illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive chemotherapy
8. Prior history of malignancy except localized basal cell, squamous skin cancer or carcinoma in situ of the cervix
9. Any prior chemotherapy or radiation therapy (except for cyclophosphamide used to treat MS disease)
10. History of sickle cell disease (SS), SC disease, coagulopathy, or if actively receiving anticoagulation therapy
11. History of insulin-dependent diabetes
12. Inability or unwillingness to pursue effective means of birth control from the time of evaluation for eligibility until 6 months post-transplant. Effective birth control is defined as (1) abstinence defined as refraining from all acts of vaginal intercourse, (2) consistent use of birth control pills, (3) injectable birth control methods (Depo-provera, Norplant), (4) tubal sterilization or male partner who has undergone vasectomy, (5) placement of an intrauterine device (IUD), or (6) with every act of intercourse, use of diaphragm with contraceptive jelly and/or use of condom with contraceptive foam
13. Failure to willingly accept or comprehend irreversible sterility as a side effect of therapy
14. Forced expiratory volume at one second (FEV1)/ forced vital capacity (FVC) < 60% of predicted after bronchodilator therapy (if necessary)
15. Diffusing capacity of the lungs for carbon monoxide (DLCO) < 60% of predicted
16. Resting left ventricular ejection fraction (LVEF) < 50 %
17. Bilirubin > 2.0 mg/dl
18. Serum creatinine > 2.0 mg/dl
19. Known hypersensitivity to mouse, rabbit, or E. Coli derived proteins or to iron compounds/medications
20. Presence of metallic objects implanted in the body that would preclude the ability of the patient to safely have MRI exams
21. Platelet count < 100,000/ul
22. White blood cell count (WBC) < 1,500 cells/mm3
23. Psychiatric illness, mental deficiency or cognitive dysfunction making compliance with treatment or informed consent impossible
24. Active infection except asymptomatic bacteriuria
25. Use of Tysabri (natalizumab) within the previous six months
26. Use of Gilenya (fingolimod) within the previous three months
27. Use of Tecfidera (dimethyl fumarate) within the previous three months
28. Use of Aubagio (teriflunomide) unless cleared from the body (plasma concentration <0.02mcg/ml) following elimination from the body with cholestyramine 8g three times a day for 11 days
29. Use of Lemtrada/Campath (alemtuzumab) within previous 12 months
30. Use of Rituxan (rituximab) or Ocrevus (ocrelizumab) within previous four months
31. Prior treatment with Novantrone (mitoxantrone)
32. Any hereditary neurological disease such as Charcot-Marie-Tooth disease (CMT), Spinocerebellar ataxia (SCA), or Parkinson's Disease
33. Severe or symptomatic cervical spinal stenosis unless surgically corrected
34. Myocardial infarction within last 12 months; if longer than 12 months, must pass dobutamine stress test and be cleared by cardiology

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- IVIg Arm: Hematopoietic Stem Cell Therapy performed as follows: Autologous stem cells will be infused after conditioning with cyclophosphamide, mesna, rATG (rabbit), and methylprednisolone. IVIg and G-CSF administered post-transplant.
  Cyclophosphamide:immunosuppressive agent;alkylating agent
  Mesna: Prophylaxis decrease for hemorrhagic cystitis
  rATG: lymphocyte-specific immunosuppressive agent which contains antibodies specific to the antigens found on the surface of T cells
  Methylprednisolone: Steroid
  G-CSF: Granulocyte-colony stimulating factor; a glycoprotein that stimulates the bone marrow to produce granulocytes & stem cells and release them into the bloodstream
  IVIg: Immunoglobulin G (IgG) products manufactured from pooled human plasma and typically contain more than 95% unmodified IgG, which has intact Fc-dependent effector functions and only trace amounts of immunoglobulin A (IgA) or immunoglobulin M (IgM).
  Autologous Stem Cells: Infusion of one's own stem cells
Period: Overall Study
Arm/Group | Control Arm | IVIg Arm
Started | 34 | 32
Completed | 33 | 31
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | IVIg Arm | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Continuous [Mean (Full Range); unit: years] | 36.3 [23 to 50] | 35.3 [20 to 48] | 35.8 [20 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 19 | 43
  Male | 10 | 13 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 28 | 28 | 56
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 34 | 32 | 66
Diagnosis of Multiple Sclerosis using revised McDonald criteria [Count of Participants; unit: Participants] | 34 | 32 | 66

OUTCOME MEASURES:

1. Primary Outcome: Efficacy - Rate of Disease Activity
Description: Defined as no relapse (defined as acute neurologic deterioration occurring after engraftment and lasting more than 24 hours, accompanied by objective worsening on neurological examination that are documented by a neurologist and not explained by fever, infection, stress, heat or related pseudoexacerbation; supportive confirmation by enhancement on MRI is preferred), no disease progression (defined as a 1.0-point increase in the Expanded Disability Status Scale (EDSS) on consecutive evaluations at least 6 months apart and not due to a non-MS disease process), and no new or enhancing lesions on MRI
Time Frame: 5 years
Population: Study Terminated due to PI taking Sabbatical: Data Not Collected
Arm/Group | Control Arm | IVIg Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 1 year post transplant
Arm/Group | Control Arm | IVIg Arm
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/31
Other Adverse Events (participants affected / at risk) | 0/33 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT03342638/Prot_002.pdf